CLINICAL TRIAL: NCT04894279
Title: A Study of the Reliability and Validity of the Turkish Version of Short Multidimensional Inventory Lifestyle Evaluation - Confinement
Brief Title: Reliability and Validity of the Turkish Version of SMİLE-C
Acronym: SMİLE-C
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: SMİLE-C
Record Dates: First submitted 2021-05-16; First posted 2021-05-20 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: Covid-19, pandemic, lifestyle
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
How the life style changed multidimensionally with home isolation in the period of COVID-19 is a new research question. Physical and social isolation, home isolation, and quarantine policies applied during epidemic periods such as SARS, MERS, Ebola have been associated with lifestyle changes (Lippi, 2019). Much of the research on the health impact of epidemics and isolation has focused on psychological issues such as stress-related symptoms and disorders and to a lesser extent social support and stress management. In contrast, the epidemic and its associated lifestyle issues during quarantine and isolation, including the impact of dietary changes, restricted physical activity, and increased indoor and screen time, are still not investigated. A limited number of studies have examined lifestyle changes during COVID-19 and previous epidemic periods. However, there is no Turkish survey that comprehensively deals with the lifestyle, the scope of which is expanding, today. The Brief Multidimensional Lifestyle Assessment Scale, which we planned to validate in our study, is a scale developed by Balanzá-Martínez et al to multi-dimensionally evaluate the lifestyle changes that occurred during the COVID-19 outbreak. It consists of 7 parts (Diet and Nutrition, Substance addiction, Physical activity, Stress management, Restorative sleep, Social support and Environmental exposure) and a total of 27 items. There are response options measured using a 4-point Likert scale. High scores indicate a healthy lifestyle (Balanzá-Martínez, 2021).

In this context, we think that adapting the Short Multidimensional Lifestyle Assessment Scale / Short Multidimensional Inventory Lifestyle Evaluation - Confinement (SMILE-C) questionnaire into Turkish will make a significant contribution to the literature.

ELIGIBILITY:
Inclusion Criteria:

Female and male participants aged 18-65, Volunteering to participate in research

Exclusion Criteria:

Inability to use a computer, tablet or mobile phone, Not answering all the questions in questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy people between 18-65 years old.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Short Multidimensional Inventory Lifestyle Evaluation - Confinement | 5 minutes
  Questionnaire
Health Promoting Life-Style Profile | 10 minutes
  Questionnaire
International Physical Activity Questionnaire - Short Form | 5 minutes
  Quesitonnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Berivan Beril KILIÇ, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Balanza-Martinez V, Kapczinski F, de Azevedo Cardoso T, Atienza-Carbonell B, Rosa AR, Mota JC, De Boni RB. The assessment of lifestyle changes during the COVID-19 pandemic using a multidimensional scale. Rev Psiquiatr Salud Ment (Engl Ed). 2021 Jan-Mar;14(1):16-26. doi: 10.1016/j.rpsm.2020.07.003. Epub 2020 Aug 29. PMID 32962948
- [Background] Firth J, Ward PB, Stubbs B. Editorial: Lifestyle Psychiatry. Front Psychiatry. 2019 Aug 26;10:597. doi: 10.3389/fpsyt.2019.00597. eCollection 2019. No abstract available. PMID 31507466
- [Background] He H, Harris L. The impact of Covid-19 pandemic on corporate social responsibility and marketing philosophy. J Bus Res. 2020 Aug;116:176-182. doi: 10.1016/j.jbusres.2020.05.030. Epub 2020 May 21. PMID 32457556
- [Background] Jiao WY, Wang LN, Liu J, Fang SF, Jiao FY, Pettoello-Mantovani M, Somekh E. Behavioral and Emotional Disorders in Children during the COVID-19 Epidemic. J Pediatr. 2020 Jun;221:264-266.e1. doi: 10.1016/j.jpeds.2020.03.013. Epub 2020 Apr 3. No abstract available. PMID 32248989
- [Background] Lippi G, Henry BM, Sanchis-Gomar F. Physical inactivity and cardiovascular disease at the time of coronavirus disease 2019 (COVID-19). Eur J Prev Cardiol. 2020 Jun;27(9):906-908. doi: 10.1177/2047487320916823. Epub 2020 Apr 9. No abstract available. PMID 32270698
- [Background] Pinar R, Celik R, Bahcecik N. Reliability and construct validity of the Health-Promoting Lifestyle Profile II in an adult Turkish population. Nurs Res. 2009 May-Jun;58(3):184-93. doi: 10.1097/NNR.0b013e31819a8248. PMID 19448522
- [Background] Orru G, Ciacchini R, Gemignani A, Conversano C. Psychological Intervention Measures During the Covid-19 Pandemic. Clin Neuropsychiatry. 2020 Apr;17(2):76-79. doi: 10.36131/CN20200208. PMID 34908972
- [Background] GBD 2017 Risk Factor Collaborators. Global, regional, and national comparative risk assessment of 84 behavioural, environmental and occupational, and metabolic risks or clusters of risks for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1923-1994. doi: 10.1016/S0140-6736(18)32225-6. Epub 2018 Nov 8. PMID 30496105
- [Background] Tabachnick, B. G., & Fidell, L. S. (2018). Using multivariate statistics (7th ed.).
- [Background] Walker, S. N., & Hill-Polerecky, D. M. (1997). Psychometric evaluation of Health Promoting Lifestyle Profile II. Unpublished manuscript, University of Nebraska Medical Center, College of Nursing, Lincoln.
- [Background] Yılmaz, Ö , Boz, H , Arslan, A . (2017). DEPRESYON ANKSİYETE STRES ÖLÇEĞİNİN(DASS 21) TÜRKÇE KISA FORMUNUN GEÇERLİLİK-GÜVENİLİRLİK ÇALIŞMASI . Finans Ekonomi ve Sosyal Araştırmalar Dergisi , 2 (2) , 78-91 . Retrieved from. https://dergipark.org.tr/tr/pub/fesa/issue/30912/323190